CLINICAL TRIAL: NCT01564095
Title: TOP-Study (Tacrolimus Organ Perfusion): A Prospective Multicenter Trial for Treatment of Ischemia Reperfusion Injury in Marginal Organs With an ex Vivo Tacrolimus Perfusion
Brief Title: TOP-Study (Tacrolimus Organ Perfusion): Treatment of Ischemia Reperfusion Injury in Marginal Organs With an ex Vivo Tacrolimus Perfusion
Acronym: TOP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Missing evidence of the effectiveness of the study medication
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. M. Angele, Prof. Dr. med. Martin Angele, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOP-Study
Record Dates: First submitted 2012-03-14; First posted 2012-03-27 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Terminal Liver Disease; Ischemia Reperfusion Injury; Graft Dysfunction; Graft Failure; Poor Graft Quality
Keywords: Liver transplantation; EDC; IRI; graft survival; graft function; graft preconditioning; Tacrolimus rinse; randomised multicenter trial
MeSH Terms: conditions — Reperfusion Injury | interventions — Tacrolimus; Receptor, EphB4

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus + HTK (Experimental): Ex vivo Tacrolimus Rinse (20 ng/ml solved in 1000 ml HTK) of marginal liver grafts prior to implantation
  Interventions: Drug: Tacrolimus
- HTK (Placebo Comparator): Ex vivo Rinse (1000 ml HTK) of marginal liver grafts prior to implantation
  Interventions: Drug: HTK/Placebo

INTERVENTIONS:
Drug: Tacrolimus — Marginal liver grafts are flushed with Tacrolimus (20ng/ml) solved in 1000 ml HTK preservation solution (duration: 15 min) ex vivo at the end of backtable preparation in the experimental group.
  Other Names: Tacrolimus, Prograf; Astellas Germany; HTK, histidin-tryptophane-ketoglurate organ preservation solution, Custodiol, Dr. Franz Köhler Chemie, Germany
  Arms: Tacrolimus + HTK
Drug: HTK/Placebo — Marginal liver grafts are flushed with 1000 ml HTK preservation solution(duration: 15 min) ex vivo at the end of backtable preparation in the placebo group.
  Other Names: HTK, histidin-tryptophane-ketoglurate organ preservation solution, Custodiol, Dr. Franz Köhler Chemie, Germany
  Arms: HTK

SUMMARY:
Utilisation of extended criteria donors due to critical organ shortage contributes to increased ischemia reperfusion injury as well as mortality following liver transplantation. Experimental data show protective effects on hepatic ischemia reperfusion injury (IRI) using the calcineurin inhibitor Tacrolimus applied intravenously or directly as a hepatic rinse. Moreover clinical data indicate a protective role of a Tacrolimus rinse in human liver transplantation when using normal, healthy grafts. The effects of Tacrolimus on hepatic injury in extended donor criteria (EDC) liver grafts remain unclear. Therefore, the aim of the present study is to examine the effects of a Tacrolimus ex vivo rinse (20 ng/ml) on cellular injury after transplantation of marginal liver grafts exhibiting 2 or more EDCs according to Eurotransplant's definition of EDC grafts.

ELIGIBILITY:
Inclusion Criteria:

Recipient:

Chronical terminal liver failure, age > 18 years, first organ transplantation

Donor:

* donor age > 65 Jahre
* macrovesicular steatosis > 40% (macroscopy or biopsy)
* BMI > 30
* sodium >165 mmol/l
* ICU stay and ventilation > 7 days
* cold ischemia time > 13 hours
* AST > 99 U/l
* ALT > 105 U/l
* bilirubin > 3 mg/dl (> 51 µmol/l)
* application of epinephrine

Exclusion Criteria:

Donor:

• Hepatitis B- or Hepatitis C-infection

Recipient:

* Multi organ transplantation
* high urgency listing
* extrahepatic tumor disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Maximum serum ALT-level | 48 hrs following liver transplantation

SECONDARY OUTCOMES:
ALT | 1,2,4,7 days after surgery
Graft survival | 7 days
AST | 1,2,4,7 days after surgery
Bilirubin | 1,2,4,7 days after surgery
Creatinin | 1,2,4,7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Angele, M.D., Principal Investigator — Ludwig-Maximilians-University, Department of Surgery, Munich, Germany; Sebastian Pratschke, M.D., Study Director — Ludwig-Maximilians-University, Department of Surgery, Munich, Germany; Karl-Walter Jauch, M.D., Study Chair — Ludwig-Maximilians-University, Department of Surgery, Munich, Germany
Locations (7):
- Germany (7):
  - Department of General, Visceral and Transplantation Surgery, Charité Campus Virchow-Klinikum, Berlin
  - Department of General and Visceral Surgery, Johann Wolfgang Goethe-University, Frankfurt am Main
  - Department of General, Visceral and Transplantation Surgery, Ruprecht Karls University, Heidelberg
  - Department of Transplantation Surgery, Johannes Gutenberg University, Mainz
  - Ludwig-Maximilians University, Campus Grosshadern, Department of Surgery, Munich
  - Department of Surgery, University of Regensburg, Regensburg
  - Department of General, Visceral and Transplantation Surgery, Eberhard Karls University, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pratschke S, Bilzer M, Grutzner U, Angele M, Tufman A, Jauch KW, Schauer RJ. Tacrolimus preconditioning of rat liver allografts impacts glutathione homeostasis and early reperfusion injury. J Surg Res. 2012 Jul;176(1):309-16. doi: 10.1016/j.jss.2011.07.045. Epub 2011 Aug 25. PMID 21962731
- [Background] St Peter SD, Post DJ, Rodriguez-Davalos MI, Douglas DD, Moss AA, Mulligan DC. Tacrolimus as a liver flush solution to ameliorate the effects of ischemia/reperfusion injury following liver transplantation. Liver Transpl. 2003 Feb;9(2):144-9. doi: 10.1053/jlts.2003.50018. PMID 12548508
- [Background] Kristo I, Wilflingseder J, Kainz A, Marschalek J, Wekerle T, Muhlbacher F, Oberbauer R, Bodingbauer M. Effect of intraportal infusion of tacrolimus on ischaemic reperfusion injury in orthotopic liver transplantation: a randomized controlled trial. Transpl Int. 2011 Sep;24(9):912-9. doi: 10.1111/j.1432-2277.2011.01284.x. Epub 2011 Jun 14. PMID 21672049
- [Result] Pratschke S, Arnold H, Zollner A, Heise M, Pascher A, Schemmer P, Scherer MN, Bauer A, Jauch KW, Werner J, Guba M, Angele MK. Results of the TOP Study: Prospectively Randomized Multicenter Trial of an Ex Vivo Tacrolimus Rinse Before Transplantation in EDC Livers. Transplant Direct. 2016 May 4;2(6):e76. doi: 10.1097/TXD.0000000000000588. eCollection 2016 Jun. PMID 27500266
- [Derived] Pratschke S, Eder M, Heise M, Nadalin S, Pascher A, Schemmer P, Scherer MN, Ulrich F, Wolters H, Jauch KW, Wohling D, Angele MK. Protocol TOP-Study (tacrolimus organ perfusion): a prospective randomized multicenter trial to reduce ischemia reperfusion injury in transplantation of marginal liver grafts with an ex vivo tacrolimus perfusion. Transplant Res. 2013 Mar 4;2(1):3. doi: 10.1186/2047-1440-2-3. PMID 23497558